CLINICAL TRIAL: NCT04648436
Title: Survival and Quality of Life After Early Surgical Intervention Versus Wait-and-see in Elderly Patients With a Traumatic Acute Subdural Hematoma (ASDH): a Pragmatic Randomized Controlled Trial With Multicenter Parallel Group Design
Brief Title: Evaluation of Surgery in Elderly With Traumatic Acute SubDural Hematoma
Acronym: RESET-ASDH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion / COVID-19 regulations
Sponsor: Leiden University Medical Center (Other)
Collaborators: Haaglanden Medisch Centrum (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Medisch Spectrum Twente (Other); Radboud Universitair Medisch Centrum (Unknown); Utrecht Universitair Medisch Centrum (Unknown); Universitair Ziekenhuis Leuven (Unknown); Algemeen Ziekenhuis Sint-Jan Brugge (Unknown); Université Libre de Bruxelles (Other); Erasme University Hospital (Other); University Hospital, Antwerp (Other); Ziekenhuis Oost-Limburg (Other); Centre Hospitalier Universitaire de Liege (Other); Algemeen Ziekenhuis Delta (Unknown); Funding agencies: ZonMw / KCE (BeNeFIT) (Unknown)
Responsible Party: Principal Investigator, wcpeul, Professor and Chair Neurosurgery, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL72116.058.20/P20.005
Record Dates: First submitted 2020-11-16; First posted 2020-12-01 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Intracranial Hemorrhages; Surgery
Keywords: Neurosurgery; Acute subdural hematoma; Traumatic brain injury
MeSH Terms: conditions — Intracranial Hemorrhages; Hematoma, Subdural, Acute; Brain Injuries, Traumatic | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with parallel group design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early surgery (Other)
  Interventions: Other: Early neurosurgical hematoma evacuation
- Initial conservative treatment (Other)
  Interventions: Other: Conservative treatment (best medical management)

INTERVENTIONS:
Other: Early neurosurgical hematoma evacuation — Early neurosurgical hematoma evacuation (preferably within 2 hours)
  Arms: Early surgery
Other: Conservative treatment (best medical management) — Conservative treatment (best medical management) on the ICU or ward
  Arms: Initial conservative treatment

SUMMARY:
Rationale: The rapidly increasing number of elderly (≥ 65 years old) with traumatic brain injury (TBI) is accompanied by substantial medical and economic consequences. An intracranial hematoma, specifically an acute subdural hematoma (ASDH), is the most common injury in elderly with TBI. The surgical versus conservative treatment of this patient group remains an important clinical and moral dilemma, since it is in most cases unclear which treatment leads to a better outcome for the patient. Current guidelines are not based on high-quality evidence and compliance is low, allowing for large treatment variation in both Belgium and the Netherlands for patients with a traumatic ASDH. In addition, elderly are underrepresented in scientific TBI literature and are therefore not included in current guidelines or prognostic models, leading to major uncertainty in (neurosurgical) decision-making for this group. As participants in two large TBI research projects (CENTER-TBI, Net-QuRe), the investigators observe that the uncertainty regarding treatment of elderly with a traumatic ASDH will not be solved by the current ongoing studies. Therefore, they recognize the necessity of undertaking a prospective, randomized, multicenter trial on the (cost-)effectiveness of early surgical hematoma evacuation versus a conservative treatment in elderly with a traumatic ASDH.

Objective: To compare the (cost-)effectiveness of early surgical hematoma evacuation versus a conservative treatment in elderly patients with a traumatic ASDH.

Study design: A prospective, pragmatic, multicenter, randomized controlled trial (RCT).

Study population: Patients ≥ 65 years with at first presentation a GCS ≥ 9 and a traumatic ASDH >10 mm or a traumatic ASDH <10 mm and a midline shift >5 mm, or a GCS < 9 with a traumatic ASDH <10 mm and a midline shift <5 mm without extracranial explanations for the comatose state, for whom clinical equipoise exists regarding the preferred treatment.

Intervention: Patients are randomized to either early surgical hematoma evacuation (A) or conservative management on the ICU or the ward (B). In case of neurological deterioration during conservative management, delayed surgery can be performed. The exact neurosurgical technique will be left to the discretion of the surgeons.

Main study parameters/endpoints: Functional outcome after 1 year, expressed by the rating on the Extended Glasgow Outcome Scale (GOS-E) Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Both treatment strategies are already used in current clinical practice as standard medical care. Therefore, there are no extra risks for patients participating in the study compared to patients outside the study. Study participation adds a minimal burden of three follow-up evaluations by visit in the first year (at 3, 6 and 12 months) and subsequent yearly evaluations by phone or postal until five years after the injury. Future elderly patients with a traumatic ASDH will benefit mostly from this study's results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* A GCS of ≥ 9 and a traumatic ASDH >10 mm in diameter or a traumatic ASDH <10 mm but with a midline shift >5 mm, or a GCS <9 and a traumatic ASDH <10 mm and a midline shift <5 mm without extracranial explanations for the comatose condition
* Clinical equipoise exists (i.e. the responsible neurosurgeon is uncertain about the benefits of either treatment)
* Informed consent is obtained or deferred

Exclusion Criteria:

* Additional epidural hematoma (EDH) or infratentorial (e.g. cerebellar) intracerebral hemorrhage (ICH)
* Major traumatic abdominal or thoracic injury (each separately defined as an Abbreviated Injury Scale (AIS) score ≥ 4) or a 'moribund' state at presentation (e.g. bilaterally absent pupillary responses)
* Known terminal condition resulting in a life expectancy of less than 1 year

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended (GOS-E) | 1 year
  scale of functional outcome ranging from 1-8 in which a higher score reflects a better recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Singh RD, van Dijck JTJM, van Essen TA, Lingsma HF, Polinder SS, Kompanje EJO, van Zwet EW, Steyerberg EW, de Ruiter GCW, Depreitere B, Peul WC. Randomized Evaluation of Surgery in Elderly with Traumatic Acute SubDural Hematoma (RESET-ASDH trial): study protocol for a pragmatic randomized controlled trial with multicenter parallel group design. Trials. 2022 Mar 29;23(1):242. doi: 10.1186/s13063-022-06184-1. PMID 35351178